CLINICAL TRIAL: NCT03734120
Title: Cryogenic Preservation of Spermatozoa : Comparative Study Between Both Dry and Liquid Phase Nitrogen Storages
Brief Title: Cryogenic Preservation of Spermatozoa
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-413
Record Dates: First submitted 2018-10-23; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Fertility; Spermatic Parameters
Keywords: Cryo preservation; Spermatic nuclear quality
MeSH Terms: interventions — Cryopreservation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- men: men undergoing routine semen analysis for infertility
  Interventions: Other: cryopreservation

INTERVENTIONS:
Other: cryopreservation — Samples were frozen with a programmable freezing unit. Each semen sample was divided into two aliquots. One aliquot was plunged into liquid nitrogen and the other was stored in dry-phase nitrogen for 3 or 6 month. Thawing was performed at room temperature

SUMMARY:
The reference technique for the conservation of gametes is storage in liquid nitrogen but new vats of nitrogen vapor (storage over liquid nitrogen) or in dry phase (storage in an insulated compartment of liquid nitrogen in a tank Liquid nitrogen) also allow the storage of flakes. The purpose of this work is to evaluate the dry-phase cryopreservation technique of liquid nitrogen compared with liquid-phase storage, depending on the duration of cryopreservation.

DETAILED DESCRIPTION:
Objective: To evaluate the effects of cryopreserved sperm in dry and liquid phase nitrogen at 3 and 6 month on sperm numeration, motility, vitality, morphology, acrosomal integrity and DNA fragmentation.

Design: Experimental study, investigator was blinded to the type of Cryopreservation.

Patient(s): Semen samples were collected from patients who came in laboratory for semen analysis

Intervention: Samples were frozen with a programmable freezing unit. Each semen sample was divided into two aliquots. One aliquot was plunged into liquid nitrogen and the other was stored in dry-phase nitrogen for 3 or 6 month. Thawing was performed at room temperature.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing routine semen analysis for infertility for reproductive medicine of university hospital in Clermont-Ferrand

Exclusion Criteria:

* women

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men undergoing routine semen analysis for infertility for reproductive medicine of university hospital in Clermont-Ferrand
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Sperm DNA integrity | at 3 months
  the spermatic DNA integrity can be quantified by TUNEL method. The result will be expressed as a percentage of fragmented DNA
Sperm DNA integrity | at 6 months
  the spermatic DNA integrity can be quantified by TUNEL method. The result will be expressed as a percentage of fragmented DNA

SECONDARY OUTCOMES:
Sperm parameter post cryopreservation | at 3 and 6 months
  The Sperm motility will be measured according to WHO recommendations
Lab parameter post cryopreservation | at 3 and 6 months
  The Sperm motility will be measured according to WHO recommendations
Spermatic DNA Compaction | at 3 and 6 months
  The spermatic DNA Compaction will be determinated by chromomycine A3 labelling (CMA3). A sperm is good when it has at least 30% of positive spermatozoa to CMA3 assay
Acrosomal integrity | at 3 and 6 months
  The acrosomal integrity will be determinated by PSA-FITC labelling.

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France